CLINICAL TRIAL: NCT05494580
Title: Pamiparib in Combination With Surufatinib in Patients With Platinum-resistant Ovarian Cancer Who Received Prior Poly (ADP-ribose) Polymerase (PARP) Inhibitors: a Multicenter, Single-arm, Phase Ib/II Trial
Brief Title: Pamiparib Plus Surufatinib in Patients With Platinum-resistant Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hutchmed (Industry)
Responsible Party: Principal Investigator, Xin Huang, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-348-01
Record Dates: First submitted 2022-07-26; First posted 2022-08-10 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Platinum-resistant Ovarian Cancer; Fallopian Tube Carcinosarcoma; Primary Peritoneal Cancer
Keywords: Ovarian cancer; PARP inhibitor; Antiangiogenic agents; Platinum-resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pamiparib; Poly A; Adenosine Diphosphate Ribose; surufatinib; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Intervention Model Description: Drug: Pamiparib Drug: Surufatinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pamiparib + Surufatinib (Phase Ib/II) (Experimental): Phase Ib:
  A dose de-escalation schedule is used in the phase Ib dose finding part. Dose Level 1 (starting dose): pamiparib 40 mg administered orally twice daily (fixed dose) and surufatinib 250 mg administered orally once daily on a 21-day treatment cycle. If ≥2/6 patients experience a dose limiting toxicity (DLT), we will de-escalate to Dose Level 2: pamiparib 40 mg administered orally twice daily (fixed dose) and surufatinib 200 mg administered orally once daily on a 21-day treatment cycle. Approximately 3-12 patients will be enrolled in phase Ib study.
  Phase II:
  The phase II part will begin once the recommended phase 2 dose (RP2D) of surufatinib have been determined in the Phase Ib in order to assess antitumor activity of pamiparib and surufatinib combination. In phase II study, pamiparib 40 mg orally twice daily and surufatinib PR2D will be administered.
  Interventions: Drug: Pamiparib; Drug: Surufatinib

INTERVENTIONS:
Drug: Pamiparib — Oral
  Other Names: Poly (ADP-ribose) polymerase (PARP) inhibitor
Drug: Surufatinib — Oral
  Other Names: Tyrosine Kinase Inhibitor

SUMMARY:
A number of studies suggest that the combination of PARP inhibitors and antiangiogenic agents produce synergistic activities. Pamiparib is a small molecule inhibitor selectivity for both PARP1 and PARP2. Surufatinib is a novel small-molecule inhibitor that simultaneously targets tumor angiogenesis (via Vascular Endothelial Growth Factor Receptor [VEGFR]1, VEGFR 2, VEGFR3 and Fibroblast Growth Factor Receptor 1 [FGFR1]) and immune evasion (via Colony Stimulating Factor 1 Receptor [CSF1R]). In this trial, we aimed to evaluate the efficacy, safety and tolerability of pamiparib in combination with surufatinib in patients with platinum-resistant ovarian cancer who received prior PARP inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form;
2. Histologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer;
3. Platinum-resistant disease, defined as progression within 6 months from completion of most recent platinum-containing therapy. Subject may have been treated with additional regimen(s) subsequent to determination of platinum resistance;
4. Patients must have received one prior PARP inhibitor therapy, and there must be a ≥ 6 month interval since treatment;
5. Female participants age 18-75 years;
6. Has measurable lesion per RECIST v1.1;
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
8. Life expectancy ≥ 3 months;
9. Patients must have normal organ and bone marrow function;
10. Women of childbearing potential should have a negative serum or urine pregnancy test prior to receiving the first dose of study treatment; and should be willing to use one acceptable contraception (i.e., oral contraceptives, condoms, intrauterine devices [IUDs]) throughout the period of taking study treatment and for at least 6 months after the last dose of study drug(s).

Exclusion Criteria:

1. Histological diagnosis of mucinous adenocarcinoma;
2. Has received prior therapy with small molecule antiangiogenic receptor tyrosine kinase inhibitors (TKIs);
3. Known or suspected allergy to any of study drugs;
4. Has clinically significant cardiovascular disease within 6 months from first dose of study intervention, including New York heart association [NYHA] class > 2, unstable angina, myocardial infarction, cardiac arrhythmia associated with hemodynamic instability (including corrected QT (QTc) interval ≥ 450 ms in men, ≥ 470 ms in female);
5. Has active ulcers, gastrointestinal perforation or obstruction;
6. Active bleeding or pathologic condition that carries a high risk of bleeding;
7. Inadequately controlled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 90 mmHg) with or without treatment;
8. Major surgery within 28 days of starting study treatment;
9. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g;
10. Uncontrolled pericardial or pleural or peritoneal effusions;
11. Has a diagnosed and/or treated additional malignancy within the last 5 years. Exceptions include in situ cervical cancer, non-melanoma skin cancer, or superficial bladder tumors that has undergone potentially curative therapy;
12. Known Human Immunodeficiency Virus (HIV) infection;
13. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis;
14. Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase Ib) | first 21 days of treatment
  MTD is defined as the highest dose level at which no more than 1 out of 6 subjects experiences a dose limiting toxicity (DLT) during the first cycles. DLT is defined as: grade 3 febrile neutropenia, grade 4 hematologic toxicities, and ≥ grade 3 non-hematologic toxicities that occurred within the first cycle of treatment with pamiparib and surufatinib.
Recommended Phase 2 dose (RP2D) (Phase Ib) | first 21 days of treatment
  Determine the RP2D of the pamiparib and surufatinib combination
Response Rate (ORR) (Phase II) | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | from the first drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD.
Duration of response (DOR) | from the first drug administration up to two years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first.
Overall survival (OS) | from the first drug administration up to 2 years
  Time from the date of first study treatment administration to the date of death due to any cause.
Safety and tolerability | up to 90 days after last study treatment administration
  Incidence, nature, and severity of adverse events graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Patient Reported Outcomes (PROs) | from the first drug administration up to two years
  Determination of changes in PROs with Functional Assessment of Cancer Therapy for patients with ovarian cancer (FACT-O) questionnaire

OTHER OUTCOMES:
Biomarkers associated with the response to pamiparib combined with surufatinib | from the first drug administration up to two years
  To identify the biomarkers, including but not limited to genomic, homologous recombination deficiency (HRD), that predict the efficacy of this study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Cetntre, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided